CLINICAL TRIAL: NCT02627404
Title: Study of the Genetic and Environmental Factors of Vulnerability in Bipolar Disorders
Acronym: GAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P111002; 2008-A01465-50 (Other: IDRCB)
Record Dates: First submitted 2015-11-13; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorders; Genetic; Biomarkers; Circadian rhythm
MeSH Terms: conditions — Bipolar Disorder | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Main module (Other): Blood sample
  Interventions: Other: Blood sample; Device: actometer

INTERVENTIONS:
Other: Blood sample — A blood sample is taken at inclusion of patients in the study to perform DNA analysis
Device: actometer — To evaluate the quality of sleep, questionnaires are completed and patients wear an actometer for 21 days. They will also complete a sleep diary

SUMMARY:
Bipolar disorder is a complex, multifactorial disorder with the intervention of genetic vulnerability factors. To help the identification of these genetic factors and to improve genotype-phenotype correlation, the identification of endophenotype through the exploration of vulnerability characteristics in unaffected first degree relatives have been recommended. For this purpose, the investigator include bipolar patients, unaffected first degree relatives and control subjects to perform genetic association studies and subphenotype analyses. In this study the investigator will focus on subgroups defined according to the existence of abnormal circadian rhythm (a major indicator of bipolar vulnerability).

Lithium is the leading treatment of bipolar disorders but prophylactic lithium response is highly variable and difficult to predict due to lack of biomarkers of response. To explore lithium response variability and to identify biomarkers of response, the investigator characterise lithium response using "ALDA" scale to conduct pharmacogenetic studies and pharmacokinetic studies of lithium extended release, in the subpopulation of patients treated with lithium. As lithium is a circadian agent, the investigator will also explore the links between lithium response and circadian phenotypes. Finally, using Li7 magnetic spectroscopy, the investigator will compare lithium brain distribution in a small sample of good and partial responders to lithium.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Bipolar I, II or Not Otherwise Specified (NOS) disorders
* Euthymic
* Age > 18
* Affiliated to the French social health care system
* Somatic state compatible with a blood test
* Informed consent signed for the study
* European

Exclusion Criteria:

* Patients major protected
* Patients adopted
* Geographical origin of grandparents unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Allele frequencies | All genotyping will be performed after 6 years

SECONDARY OUTCOMES:
Mean Activity (movement per minute) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Total time in bed (minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Total time in bed with and without sleep (minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Day to day Stability in Time to bed (ratio of minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Day to day Stability in activity (ratio of minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Sleep latency (minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Total time awaken during the night (minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Time awaken during the night (minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Percentage of time sleeping (%) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Fragmentation index (ratio) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Total sleep time (minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Activity during sleep (movement per minute) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Total activity amplitude (movement per minute) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Start L5: start of the 5 hours with the lowest activity period (hours:minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Start M10: start of the 10 hours with the highest activity period (hours:minutes) | End of participation of the activity tracking module : Day 21
  Variable recorded in the activity tracking module
Plasma and erythrocyte lithium concentration (Meq/L) at different times after inclusion | At inclusion : time 0, 1 hour, 4 hours and 8 hours - At Day 30 : Time 0 and 1 hour
Lithium brain distribution using Li7 magnetic spectroscopy | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Paris, France

REFERENCES:
- [Derived] Hennion V, Scott J, Martinot V, Benizri C, Marie-Claire C, Bellivier F, Etain B. Associations between actigraphy estimates of sleep and circadian rhythmicity and psychotropic medications in bipolar disorders: An exploratory study. J Affect Disord. 2024 Mar 1;348:224-228. doi: 10.1016/j.jad.2023.12.075. Epub 2023 Dec 29. PMID 38159652
- [Derived] Loftus J, Scott J, Vorspan F, Icick R, Henry C, Gard S, Kahn JP, Leboyer M, Bellivier F, Etain B. Psychiatric comorbidities in bipolar disorders: An examination of the prevalence and chronology of onset according to sex and bipolar subtype. J Affect Disord. 2020 Apr 15;267:258-263. doi: 10.1016/j.jad.2020.02.035. Epub 2020 Feb 19. PMID 32217226
- [Derived] Geoffroy PA, Micoulaud Franchi JA, Maruani J, Philip P, Boudebesse C, Benizri C, Yeim S, Benard V, Brochard H, Leboyer M, Bellivier F, Etain B. Clinical characteristics of obstructive sleep apnea in bipolar disorders. J Affect Disord. 2019 Feb 15;245:1-7. doi: 10.1016/j.jad.2018.10.096. Epub 2018 Oct 9. PMID 30359809
- [Derived] Richard-Lepouriel H, Kung AL, Hasler R, Bellivier F, Prada P, Gard S, Ardu S, Kahn JP, Dayer A, Henry C, Aubry JM, Leboyer M, Perroud N, Etain B. Impulsivity and its association with childhood trauma experiences across bipolar disorder, attention deficit hyperactivity disorder and borderline personality disorder. J Affect Disord. 2019 Feb 1;244:33-41. doi: 10.1016/j.jad.2018.07.060. Epub 2018 Aug 6. PMID 30336349